CLINICAL TRIAL: NCT06893432
Title: Cognitive Function and Electroencephalogram Brain Network Remodeling Among Users of Hearing Aids With Age-Related Hearing Loss
Brief Title: Cognitive Function and EEG Brain Network Remodeling Among Users of Hearing Aids With ARHL
Acronym: EEG/ARHL
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-938-01
Record Dates: First submitted 2025-02-17; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-11

CONDITIONS: Age-related Hearing Loss; Age-related Cognitive Decline; Depression; Sleep Disturbance
Keywords: age-related hearing loss; cognition; electroencephalogram
MeSH Terms: conditions — Presbycusis; Depression; Parasomnias | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aided: Participants who have regularly used hearing aid(s) to improve hearing during the past six-month period.
  Interventions: Device: hearing aids
- Control: Participants without any experience of using hearing aids.

INTERVENTIONS:
Device: hearing aids — Hearing aids are a common intervention method used to address age-related hearing loss, providing amplified sound to improve hearing clarity and communication abilities for elderly individuals.
  Groups: Aided

SUMMARY:
This study intends to retrospectively collect and analyze the case data of patients with age-related hearing loss who were admitted to the Otolaryngology Department of Sun Yat-sen Memorial Hospital from January 2020 to June 2024. Participants were divided into an Aided Group and a Control Group based on whether they had regularly used hearing aids in the past six months.

Audiological, cognitive, emotional, and sleep assessments, as well as resting state electroencephalogram (EEG) features, are supposed to be compared between the two groups.

DETAILED DESCRIPTION:
This study intends to retrospectively collect and analyze the case data of patients with age-related hearing loss who were admitted to the Otolaryngology Department of Sun Yat-sen Memorial Hospital from January 2020 to June 2024. Participants were divided into an Aided Group and a Control Group based on whether they had regularly used hearing aids in the past six months.

The audiological assessment comprises pure tone audiometry, speech recognition audiometry, and sound field audiometry. The cognitive assessment includes the Mandarin version of the Montreal Cognitive Assessment (MoCA) and the Mini-Mental State Examination (MMSE). The emotional assessment consists of the 24-item Hamilton Depression Scale (HAMD) and the 15-item Geriatric Depression Scale (GDS). Sleep assessment is conducted using the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ARHL
* Aged between 50 and 90
* Complete measuring data; including pure tone audiometry, speech audiometry, cognitive screening scales and resting-state electroencephalography
* Right-handed
* Regular daily use of hearing aid(s) for six-month period prior to the test date, or no hearing aid experience

Exclusion Criteria:

* Outer/middle ear abnormalities or any other central nervous system disorders

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, we retrospectively collect clinical data of patients with ARHL who have attended the Otolaryngology Department of Sun Yat-sen Memorial Hospital from January 2020 to June 2024. All participants are native speakers of Mandarin Chinese or Cantonese (Guangdong, China). Candidates will be excluded for outer/middle ear abnormalities or any other central nervous system disorders. Thereafter, all participants were grouped depending on whether they have regularly used hearing aid(s) to improve hearing during the past six-month period.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
better-ear pure-tone averages (BEPTA) | Day1
  The pure-tone thresholds were tested using a Piano Plus diagnostic audiometer (Inventis, Italy), following the standard Hughson-Westlake method (i.e., up 5 and down 10 dB HL). Subsequently, the pure tone average (PTA) of air conduction thresholds between 500 and 4000 Hz was calculated ear by ear. Better-ear PTA of each participant will be collected for further analysis.
binaural averaged pure-tone averages (BAPTA) | Day1
  The pure-tone thresholds were tested using a Piano Plus diagnostic audiometer (Inventis, Italy), following the standard Hughson-Westlake method (i.e., up 5 and down 10 dB HL). Subsequently, the pure tone average (PTA) of air conduction thresholds between 500 and 4000 Hz was calculated ear by ear. binaural averaged PTA of each participant will be collected for further analysis.
better-ear speech recognition thresholds (BESRT) | Day1
  Speech recognition audiometry was tested using a Piano Plus diagnostic audiometer and a Chinese disyllabic version of speech material. The correct recognition rate at each 10 dB step of test intensity was recorded, covering the full range from 0% to 100% as much as possible. However, the intensity would cease increasing when it reached the maximum tolerable limit for the participant or the maximum output of the equipment. Specifically, speech recognition threshold (SRT) was defined as the signal intensity required for the test ear to achieve a 50% correct recognition rate. Better-ear SRT of each participant will be collected for further analysis.
binaural averaged speech recognition thresholds (BASRT) | Day1
  Speech recognition audiometry was tested using a Piano Plus diagnostic audiometer and a Chinese disyllabic version of speech material. The correct recognition rate at each 10 dB step of test intensity was recorded, covering the full range from 0% to 100% as much as possible. However, the intensity would cease increasing when it reached the maximum tolerable limit for the participant or the maximum output of the equipment. Specifically, speech recognition threshold (SRT) was defined as the signal intensity required for the test ear to achieve a 50% correct recognition rate. binaural averaged SRT of each participant will be collected for further analysis.
The global and subscores of the Mandarin version of the Montreal Cognitive Assessment (MoCA) | Day1
  MoCA consists of seven subcomponents, namely visual-spatial function, naming, attention, language, abstraction, delayed recall, and orientation. It scores based on whether participants answer each item correctly, with a total score of 30. A higher score indicates better cognitive function.
The global and subscores of the Mandarin version of the Mini-Mental State Examination (MMSE) | Day1
  MMSE comprises six components: temporal orientation, spatial orientation, immediate memory, attention and calculation abilities, delayed memory, and language ability. Depending on participants' accuracy in answering each test item, MMSE is scored out of 30 points. A higher score indicates better cognitive function.

SECONDARY OUTCOMES:
better-ear PTA in the aided condition (BEPTA-A) | Day1
  For the aided group, participants additionally underwent a sound field audiometry (hearing thresholds ) with their hearing aid(s) on.
  The stimuli were presented through two binaural speakers placed one meter from the participants at 45° azimuth via a Piano Plus diagnostic audiometer. During the test session, participants were seated in an upright position to ensure the height of the microphone(s) on their hearing aid(s) was consistent with the height of the geometric center of the speaker(s). Similarly, their better-ear PTA (BEPTA-A) in the aided condition will be collected for further analysis.
binaural averaged PTA in the aided condition (BAPTA-A) | Day1
  For the aided group, participants additionally underwent a sound field audiometry (hearing thresholds ) with their hearing aid(s) on.
  The stimuli were presented through two binaural speakers placed one meter from the participants at 45° azimuth via a Piano Plus diagnostic audiometer. During the test session, participants were seated in an upright position to ensure the height of the microphone(s) on their hearing aid(s) was consistent with the height of the geometric center of the speaker(s). Similarly, their binaural averaged PTA (BAPTA-A) in the aided condition will be collected for further analysis.
better-ear SRT in the aided condition (BESRT-A) | Day1
  For the aided group, participants additionally underwent a sound field audiometry (hearing thresholds ) with their hearing aid(s) on.
  The stimuli were presented through two binaural speakers placed one meter from the participants at 45° azimuth via a Piano Plus diagnostic audiometer. During the test session, participants were seated in an upright position to ensure the height of the microphone(s) on their hearing aid(s) was consistent with the height of the geometric center of the speaker(s). Similarly, their better-ear SRT (BESRT-A) in the aided condition will be collected for further analysis.
binaural averaged SRT in the aided condition (BASRT-A) | Day1
  For the aided group, participants additionally underwent a sound field audiometry (hearing thresholds ) with their hearing aid(s) on.
  The stimuli were presented through two binaural speakers placed one meter from the participants at 45° azimuth via a Piano Plus diagnostic audiometer. During the test session, participants were seated in an upright position to ensure the height of the microphone(s) on their hearing aid(s) was consistent with the height of the geometric center of the speaker(s). Similarly, their binaural averaged SRT (BASRT-A) in the aided condition will be collected for further analysis.
the global score of Pittsburgh sleep quality index (PSQI) | Day1
  PSQI scale was compiled by Buysse et al in 1989 to assess the sleep quality of individuals in the last 1 month. The total score ranges from 0 to 21. A higher score indicates worse sleep quality in the past month.
the global score of Hamilton Depression Scale -24 items (HAMD-24) | Day1
  The HAMD-24 was used to assess the degree of depression and emotional state in patients with chronic subjective tinnitus. The assessment included the emotional state and symptoms of autonomic nervous system disorders in the past week, and each question was scored according to the presence and severity of symptoms. The total score ranges from 0 to 76. A higher score indicates worse emotion state in the past week.
the global score of 15-item Geriatric Depression Scale (GDS-15) | Day1
  GDS-15 is a self-rated depression questionnaire, with higher scores indicating a worse depressive state. The total score ranges from 0 to 15. A higher score indicates worse emotion state in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Haidi Yang, Prof., Study Director — SunYatSunU2H
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong 510000, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No